CLINICAL TRIAL: NCT04345549
Title: Ayurveda Self-Management for Flu Like Symptoms in People Self-Isolated for 7 Days During the Coronavirus Disease 2019 (COVID-19) Outbreak
Brief Title: Ayurveda Self-Management for Flu Like Symptoms During the Covid-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU08
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Flu Like Symptom; Flu Like Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda (Experimental): All the participants were advised to self-isolate for 7-days and maintain hygiene and self-care as per recommended guidelines. Along with that, participants were advised to constitution based Ayurveda treatment using herbs, life style and yoga.
  Interventions: Other: Individualised Ayurveda

INTERVENTIONS:
Other: Individualised Ayurveda — Saline warm water gargle, Steam, Paracetamol for body temperature and plenty fluid and rest, Food and herbs recommendation as per individual Ayurveda constitution, Using Ginger/ lemon/ turmeric/ honey recommended as per individual, Yoga breathing

SUMMARY:
From the end of January 2020, Coronavirus disease 2019 began to spread in United Kingdom (UK). During the same time, seasonal flu continued to circulate across the UK. With similar course of management at early stages, flu like symptoms were self-isolated to prevent the spread and further complications of infection. Present study aimed to evaluate the effect of self-managed Ayurveda on flu like symptoms in people who self-isolated at home for 7-days in March 2020 during the Covid-19 outbreak in UK.

ELIGIBILITY:
Inclusion Criteria:

* Flu like symptoms present at least one respiratory symptom (e.g. cough, nasal obstruction, sore throat) and at least one constitutional symptom other than fever (e.g. fatigue, headache, myalgias) of less than 48-hour duration
* Willing to consent and follow up

Exclusion Criteria:

* Pregnant/lactating
* Participants with chronic pulmonary diseases or critical condition or already developed severe respiratory distress
* Clinically malignancies, systemic infection, other medical or psychiatric condition which places the subject at unacceptable risk to participate in the study - Known hypersensitivity to any ayurveda herbal substances

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Time to achieve afebrile | From Baseline to 3rd and 7th-days of intervention
  Time to bring down a fever (oral temperature < 37.2˚C)

SECONDARY OUTCOMES:
Severity of influenza symptom score | Twice daily from Day 1 to Day 7
  Symptoms diary card completed twice daily from Day 0 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Principal Investigator — Aarogyam UK; Jaydeep Joshi, Study Director — Aarogyam UK
Locations (1):
- Aarogyam, Leicester, United Kingdom